CLINICAL TRIAL: NCT05482789
Title: Pilot Study of Exenatide Pharmacokinetics and Pharmacodynamics in Gestational Diabetes
Brief Title: Exenatide Pharmacokinetics and Pharmacodynamics in Gestational Diabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Maisa N. Feghali, MD (Other)
Responsible Party: Sponsor-Investigator, Maisa N. Feghali, MD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY22070080
Record Dates: First submitted 2022-07-18; First posted 2022-08-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Exenatide (Experimental): Participant receives injection of 10 micrograms of Exenatide sub-cutaneously the given mixed meal test and blood samples will be drawn for laboratory testing.
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — 10 microgram injected sub-cutaneously once

SUMMARY:
This study is being done to study how exenatide, an FDA-approved drug that lowers blood sugar in non-pregnant patients with type II diabetes, works in pregnant women. To do this, the investigators will study the drug's pharmacokinetics (what the body does to the drug; specifically, how quickly your body breaks down and excretes exenatide) and pharmacodynamics (what the drug does to the body; specifically, how effectively exenatide helps the participants' pancreas secrete insulin and how well it controls blood sugar after a meal). There are only two main drug therapies (insulin injections and glyburide pills) currently used for gestational diabetes and not all women achieve good enough blood sugar control without side effects. Therefore, the investigators hope to find out if exenatide might also be helpful in gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (singleton)
* Gestational diabetes not requiring medical therapy
* Between 18 and 50 years of age
* Able to give written informed consent

Exclusion Criteria:

* Women in the first trimester of pregnancy
* Hematocrit less than 30%
* Current or past treatment with any hypoglycemic agent
* Women with gastrointestinal disease or symptoms consistent with nausea, vomiting, abdominal pain or reflux requiring medical treatment.
* Women with high triglyceride levels, history of gallbladder or pancreatic disease.
* Clinical diagnosis or history of any renal insufficiency (or decreased creatinine clearance)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) of glucose | Baseline and 1 week later
  Glucose concentration over the course of each study visit following mixed tolerance test

SECONDARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) of exenatide | 1 week after study enrollment
  Drug concentration over the course of the second study visit

CONTACTS AND LOCATIONS:
Overall Officials: Maisa Feghali, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No